CLINICAL TRIAL: NCT01083394
Title: Randomized Trial of Paclitaxel Eluting Balloon or Conventional Balloon for Treatment of In-Stent Restenosis of the Superficial Femoral Artery in Patients With Symptomatic Peripheral Artery Disease (ISAR-PEBIS)
Brief Title: Paclitaxel Eluting Balloon and Conventional Balloon for In-Stent Restenosis of the Superficial Femoral Artery
Acronym: ISAR-PEBIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE IDE No. B00210
Record Dates: First submitted 2010-02-26; First posted 2010-03-09 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2010-04

CONDITIONS: Peripheral Vascular Disease
Keywords: PTA; paclitaxel; restenosis
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional PTA (Active Comparator): In stent restenosis is treated with PTA using a conventional balloon.
  Interventions: Device: PTA; Procedure: Percutaneous Transluminal Angioplasty (PTA)
- PTA with PEB (Experimental): In stent restenosis is treated with PTA using a paclitaxel eluting balloon.
  Interventions: Device: PTA with PEB; Procedure: Percutaneous Transluminal Angioplasty (PTA)

INTERVENTIONS:
Device: PTA — PTA using a conventional balloon
  Other Names: PACIFIC XTREME, Invatec
  Arms: conventional PTA
Device: PTA with PEB — PTA using a paclitaxel eluting balloon
  Other Names: IN.PACT PACIFIC, Invatec
  Arms: PTA with PEB
Procedure: Percutaneous Transluminal Angioplasty (PTA) — Percutaneous transluminal angioplasty with conventional balloon or paclitaxel-eluting balloon
  Other Names: PACIFIC XTREME or IN.PACT PACIFIC balloons

SUMMARY:
The aim of this study is to perform a randomized, controlled trial to compare percutaneous transluminal angioplasty using paclitaxel eluting balloon (PEB) or using a conventional balloon for treatment of superficial femoral artery in-stent restenosis.

DETAILED DESCRIPTION:
The superficial femoral artery is a common place for arteriosclerosis in patients symptomatic for lower extremity vascular disease. Advances in percutaneous transluminal angioplasty (PTA) and stenting have provided new options for the treatment of the disease in this arterial segment. Restenosis after PTA occurs in 40-60% within one year. A novel attempt to reduce restenosis is the use of paclitaxel eluting balloons (PEB). First clinical studies suggest that the use of PEBs during percutaneous treatment of femoropopliteal disease is associated with significant reductions in late lumen loss and target-lesion revascularization. There is no randomized comparison of these treatments in patients with in stent restenosis of the superficial femoral artery. Thus, the aim of this study was to compare the efficacy of PTA with conventional balloon or PEB for in stent restenosis in the SFA in terms of reduction of diameter stenosis at follow-up angiogram.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic ≥ 70% in-stent restenosis of the AFS, (Rutherford stage 2-6)
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study

Exclusion Criteria:

* Acute ischemia and/or acute thrombosis of the SFA
* Untreated ipsilateral iliac artery stenosis >70%
* Not at least one vessel run-off
* Popliteal involvement with stenosis >70%
* Severe renal insufficiency (GFR <30 ml/min/m2)
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Previous enrollment in this trial.
* Patient's inability to fully cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Percentage diameter stenosis | 6 months

SECONDARY OUTCOMES:
All-cause mortality | 6 and 24 months
Major adverse peripheral events (MAPE) defined as acute thrombosis of SFA or ipsilateral amputation or revascularization (PTA or bypass surgery) | 6 Months
Time to onset of any of MAPE | 3-24 months
Binary restenosis rate | 6 months
Percentage diameter stenosis in duplex ultrasound | 6 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum Muenchen; Ilka V. Ott, MD, Principal Investigator — Klinikum rechts der Isar
Locations (2):
- Germany (2):
  - 1. Medizinische Klinik, Klinikum rechts der Isar, München
  - Deutsches Herzzentrum, München

REFERENCES:
- [Derived] Ott I, Cassese S, Groha P, Steppich B, Voll F, Hadamitzky M, Ibrahim T, Kufner S, Dewitz K, Wittmann T, Kasel AM, Laugwitz KL, Schunkert H, Kastrati A, Fusaro M. ISAR-PEBIS (Paclitaxel-Eluting Balloon Versus Conventional Balloon Angioplasty for In-Stent Restenosis of Superficial Femoral Artery): A Randomized Trial. J Am Heart Assoc. 2017 Jul 25;6(7):e006321. doi: 10.1161/JAHA.117.006321. PMID 28743787